CLINICAL TRIAL: NCT04263350
Title: An Open-label, Randomized Crossover Study to Obtain a Preliminary Estimate of the Bioavailability of Atazanavir and Cobicistat When Administered in an Age-appropriate Fixed-Dose Combination Formulation Compared With Coadministration of the Age-appropriate Atazanavir and Cobicistat Individual Formulations and to Assess Preliminary Palatability/Acceptability in Healthy Adults
Brief Title: A Study to Examine the Acceptable Taste and to Estimate the Amount of Atazanavir and Cobicistat in the Body When Taken as a Combination Product Versus When Taken as Separate Products at the Same Time
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AI424-567
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Healthy Participants
Keywords: Healthy Participants
MeSH Terms: interventions — Atazanavir Sulfate; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A:Fixed- dose combination mini-tablet (Experimental)
  Interventions: Drug: Atazanavir/Cobicistat
- Treatment B: Separate products taken at the same time (Experimental)
  Interventions: Drug: Reyataz Atazanavir; Drug: Cobicistat

INTERVENTIONS:
Drug: Atazanavir/Cobicistat — Specified Dose on Specified Days
  Other Names: ATV/COBI
  Arms: Treatment A:Fixed- dose combination mini-tablet
Drug: Reyataz Atazanavir — Specified Dose on Specified Days
  Other Names: REYATAZ (ATV)
  Arms: Treatment B: Separate products taken at the same time
Drug: Cobicistat — Specified Dose on Specified Days
  Other Names: COBI
  Arms: Treatment B: Separate products taken at the same time

SUMMARY:
The purpose of this study is to compare the amount of Atazanavir (ATV) and Cobicistat (COBI) in the bodies of healthy adult participants when taken as a combination formulation, and when ATV is administered as an oral powder at the same time as COBI administered as an oral tablet. The ATV/COBI combination formulation and ATV powder will be taken with food.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive.
* Women and men must agree to follow specific methods of contraception, if applicable.

Exclusion Criteria:

* History of a clinically significant drug rash or Stevens-Johnson Syndrome
* History of Gilbert's Syndrome
* Current or recent (within 3 months of administration) gastrointestinal disease that could impact upon the absorption of study treatment
* Any major surgery within 4 weeks of study treatment administration
* Any gastrointestinal surgery that could impact upon the absorption of study treatment

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Atazanavir (ATV) | Up to Day 10
Cmax of Cobicistat (COBI) | Up to Day 10
Area under the plasma concentration- time Curve from time zero extrapolated to infinite time (AUC(INF)) of ATV | Up to Day 10
AUC(INF) of COBI | Up to Day 10

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Up to 70 days
Incidence of AEs leading to discontinuation | Up to 40 days
Incidence of deaths | Up to 40 days
Marked abnormalities in clinical laboratory test results | Up to 40 days
Incidence of marked abnormalities in vital sign measurements: Blood Pressure | Up to 40 days
Incidence of marked abnormalities in vital sign measurements: Heart Rate | Up to 40 days
Incidence of marked abnormalities in Electrocardiogram (ECG) recording | Up to 40 days
Incidence of Palatability questionnaire results | Up to 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm